CLINICAL TRIAL: NCT02324660
Title: Prospective Evaluation of a Screening Methodology for Chronic Obstructive Pulmonary Disease in Patients Admitted to Hospital for Acute Coronary Syndromes.
Brief Title: Screening for Chronic Obstructive Pulmonary Disease in Patients With Acute Coronary Syndromes
Acronym: SCAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital of Ferrara (Other)
Responsible Party: Principal Investigator, Gianluca Campo, MD, University Hospital of Ferrara
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 131295
Record Dates: First submitted 2014-12-18; First posted 2014-12-24 (Estimated); Results first posted 2017-08-07 (Actual); Last update posted 2017-08-07 (Actual); Status verified 2017-05

CONDITIONS: Chronic Obstructive Pulmonary Disease; Acute Coronary Syndromes
Keywords: screening procedure; peak expiratory flow; respiratory health screening questionnaire
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Acute Coronary Syndrome | interventions — Mass Screening

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- screening test (Other): all consecutive patients admitted to our hospital for ACS and current/former smokers will be screened according our protocol with PEF and RHSQ. Patients will be blinded to result of both tests. Indipendently to results, all included patients will receive spirometry (50-70 days after inclusion) to assess the presence or not of COPD (primary outcome).
  Interventions: Other: screening test

INTERVENTIONS:
Other: screening test — screening test with peak expiratory flow and respiratory health screening questionnaire to discriminate patients at risk for COPD

SUMMARY:
Several studies and registries suggested that the concomitant presence of acute coronary syndromes (ACS) and chronic obstructive pulmonary disease (COPD) is significantly associated with poor prognosis. It has been suggested that diagnosis of COPD is frequently missing. Thus, it is plausible that a significant percentage of patients with ACS may have unrecognized COPD. This missing diagnosis may contribute significantly to poor prognosis. The investigators suppose that the concomitant use of peak expiratory flow (PEF) measurement and of Respiratory Health Screening Questionnaire (RHSQ, adapted version) could be useful as screening test for COPD in patient smokers or former smokers admitted to hospital with a diagnosis of ACS. In all screened patients COPD diagnosis will be confirmed (or not) two months after hospital discharge with spirometry. In the same setting of patients, the investigators will characterize the underlying pathological mechanisms, evaluating several inflammation, platelet and endothelial markers.

DETAILED DESCRIPTION:
BACKGROUND:

Acute coronary syndromes (ACS) and chronic obstructive pulmonary disease (COPD) are respectively the first and the fourth leading cause of death in Western countries. ACS and COPD shared several risk factor, in particular smoking habitus. Available data may be summarized as follows: i) ACS, and generally ischemic heart disease (IHD), are the most frequent comorbidity in COPD patients; ii) cardiac adverse events are the most frequent cause of hospitalization and/or death in COPD patients; iii) patients with ACS and concomitant COPD are at higher risk of mortality, re-infarction and heart failure (HF); iv) COPD is frequently undiagnosed in patients with IHD. At the best of our knowledge, no studies investigated the effectiveness and feasibility of screening procedures to early detect COPD in ACS patients. The identification of unrecognized COPD in ACS patients may permit an optimization of the treatment with an significant improvement in the outcome. Finally, it is well known that several biological processes are involved in the development and worsening of IHD-COPD comorbidity (e.g. inflammation, hypoxia, heightened platelet reactivity, endothelial dysfunction). Nevertheless, a complete evaluation of these processes is currently missing. A better characterization of these biological processes underlying the ACS-COPD comorbidity may significantly improve its management.

HYPOTHESIS and SIGNIFICANCE:

Based on previous studies in patients with stable IHD, we suppose that at least 30% of patients admitted to hospital for ACS have undiagnosed COPD. They represent a subgroup of patients at very high risk of death, reinfarction and heart failure. We hypothesize that the combined use of PEF and RHSQ (adapted version) in ACS patients (smokers or former smokers) before hospital discharge may discriminate those with undiagnosed COPD. The early diagnosis of COPD comorbidity may have important clinical implications. We speculate that early identification of undiagnosed COPD in ACS patients may permit a promptly treatment and improve outcomes. Finally, we suppose that the worst outcome observed in ACS patients with undiagnosed COPD as well as in patients with prior ACS and acute exacerbation of COPD is due to a specific pattern of alterations in platelet reactivity (PR), endothelial function (EF) and inflammation. Therefore, their characterization may lead to an improvement in the clinical management of these patients.

METHODS:

Blood samples: At the time of enrollment an aliquot (7-10 ml) of whole blood will be collected and stored for DNA and RNA extraction. Blood samples to obtain plasma (7-10 ml) and serum (7-10 ml) will be collected both at the timing of enrolment and at the time of spirometry.

Screening procedure: PEF and RHSQ (adapted version) will be administered by an independent combined team of cardiologist and pulmonologist before the hospital discharge. According to international guidelines, patients will be asked to perform 3 consecutive PEF measurements and the highest values will be recorded. A PEF value below 80% predicted will be considered predictive of impaired lung function. The RHSQ questionnaire will be performed as previously reported with a value >19 suggesting high probability of COPD.

Spirometry: spirometry test will be performed 50-70 days after hospital discharge (enrollment time).

Primary outcome of the study: the endpoint of the study is the diagnosis of COPD at spirometry. The aim of the study is to establish if the combined use of PEF and RHSQ questionnaire is able to early predict COPD diagnosis.

Clinical follow-up: a complete 1-year follow-up will be collected in each patient recording the occurrence of all adverse events and hospital admissions. All adverse events will be adjudicated by two independent reviewers blinded to screening and spirometry outcomes.

Biological parameters: several evaluations of inflammation, endothelial and platelet function markers will be performed in blood samples from patients. The principals are reported below: high sensitivity C-reactive protein, fibrinogen, interleukin (IL)-6, IL-1Ra, tumor necrosis factor (TNF)-alpha, platelet reactivity as assessed by light transmission aggregometry and VerifyNow system, ICAM and Bcl-2 and e-NOS (extracellular nitric oxide synthase) (in human umbilical vein endothelial cells that will be incubate with serum of patients), intracellular levels of reactive oxygen species.

Secondary outcomes: PEF, RHSQ, biological parameters and spirometry results will be related to clinical outcome.

ELIGIBILITY:
Inclusion Criteria:

* age >40 years
* typical chest pain during at least 20 minutes
* ST-segment changes on electrocardiography, indicating ischemia and/or positive test of a biomarker (troponin and/or CK-MB), indicating myocardial necrosis
* current or former history of smoking

Exclusion Criteria:

* previous diagnosis of COPD and/or asthma
* known pulmonary disease
* ongoing pneumonia
* ongoing heart failure
* documented or suspicion of malignant disease
* life expectancy <1 year
* recent thoracic trauma

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 137 (Actual)
Dates: Start 2014-12; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gianluca Campo, MD, Principal Investigator — University Hospital of Ferrara; Marco Contoli, MD, Principal Investigator — University Hospital of Ferrara
Locations (1):
- University Hospital of Ferrara, Cona, Ferrara, Italy

REFERENCES:
- [Result] Campo G, Pavasini R, Barbetta C, Maietti E, Mascetti S, Biscaglia S, Zaraket F, Spitaleri G, Gallo F, Tonet E, Papi A, Ferrari R, Contoli M. Predischarge screening for chronic obstructive pulmonary disease in patients with acute coronary syndrome and smoking history. Int J Cardiol. 2016 Nov 1;222:806-812. doi: 10.1016/j.ijcard.2016.08.030. Epub 2016 Aug 4. PMID 27522379
- [Derived] Erriquez A, Pavasini R, Biscaglia S, Tebaldi M, Tonet E, Maietti E, Cimaglia P, Grazzi G, Scoccia A, Cardelli LS, Verardi FM, Morelli C, Campana R, Rubboli A, Mazzoni G, Volpato S, Ferrari R, Campo G. The impact of periprocedural myocardial infarction on mortality in older adults with non-ST-segment elevation acute coronary syndrome: a pooled analysis of the FRASER and HULK studies. J Cardiovasc Med (Hagerstown). 2021 Jul 1;22(7):546-552. doi: 10.2459/JCM.0000000000001146. PMID 34076602
- [Derived] Pavasini R, Fiorencis A, Tonet E, Gaudenzi E, Balla C, Maietti E, Biscaglia S, Papi A, Ferrari R, Contoli M, Campo G. Right Ventricle Function in Patients with Acute Coronary Syndrome and Concomitant Undiagnosed Chronic Obstructive Pulmonary Disease. COPD. 2019 Aug;16(3-4):284-291. doi: 10.1080/15412555.2019.1645105. Epub 2019 Jul 29. PMID 31357891
- [Derived] Pavasini R, Vieceli Dalla Sega F, Gallo F, Passarini G, Papi A, Contoli M, Campo G. Endothelial dysfunction and increased platelet reactivity in patients with acute coronary syndrome and undiagnosed COPD: insights into the SCAP trial. Eur Respir J. 2017 Oct 5;50(4):1701183. doi: 10.1183/13993003.01183-2017. Print 2017 Oct. No abstract available. PMID 28982765

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From December 2014 to August 2015, 169 acute cornary syndromes patients with smoking history underwent screening procedure in the University Hospital of Ferrara
Groups:
- Patients Undergoing Screening and Spirometry: From December 2014 to August 2015, 169 ACS patients with smoking history underwent screening procedure. Screening procedure combined peak expiratory flow rate (PEFR, defined as positive if <80% of predicted) and respiratory health status questionnaire (RHSQ, defined as positive if >19.5 points). Overall, 137 (81%) patients received spirometry (final study population)
Period: Overall Study
Arm/Group | Patients Undergoing Screening and Spirometry
Started | 169
Completed | 137
Not Completed | 32

BASELINE CHARACTERISTICS:
Arm/Group | Patients Undergoing Screening and Spirometry
Number analyzed (Participants) | 137
Age, Continuous [Mean (Standard Deviation); unit: years] | 65 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 115
Region of Enrollment [Number; unit: participants]
  Italy | 137

OUTCOME MEASURES:

1. Primary Outcome: COPD Diagnosis
Description: COPD diagnosis confirmed by spirometry
Time Frame: 2 months after inclusion
Measure: Number; unit: participants
Arm/Group | Patients Undergoing Screening and Spirometry
Number analyzed (Participants) | 137
participants | 39

2. Secondary Outcome: Cardiac Adverse Events
Description: cumulative occurrence of death, myocardial infarction and heart failure
Time Frame: 1 year after inclusion
Measure: Number; unit: partecipants
Arm/Group | Screening Test
Number analyzed (Participants) | 137
partecipants | 8

3. Secondary Outcome: Undiagnosed COPD
Description: percentage of patients admitted to hospital for ACS and with undiagnosed COPD
Time Frame: 2 months
Reporting Status: Not Posted

4. Other Pre Specified Outcome: Adverse Events
Description: hospital admission for ACS, for bleeding complications, for respiratory failure, for arrhytmias, for pneumonia
Time Frame: 1 year after inclusion
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Cardiac Death
Description: occurrence of cardiac death
Time Frame: 1 year
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 2 months
Arm/Group | Patients Undergoing Screening and Spirometry
Serious Adverse Events (participants affected / at risk) | 0/137
Other Adverse Events (participants affected / at risk) | 0/137

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes